CLINICAL TRIAL: NCT05671731
Title: The Effect of Combining Prebiotic Treatment With a Diet/Physical Activity Educational Program on Body Composition and Intestinal Microbiota in 4th and 5th Grade Children
Brief Title: Combining Prebiotic and Diet/Physical Activity Educational Program Effects on Body Composition and Intestinal Microbiota in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marquette University (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2411
Record Dates: First submitted 2022-12-20; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Obesity, Childhood
Keywords: prebiotics; Gastrointestinal Microbiome; Hispanic or Latino
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: cluster randomized controlled feasibility trial
Who Masked: Outcomes Assessor
Masking Description: Research assistants collecting data did not know group assignment of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group received Beneo Synergy 1 - 4gm twice/school day in 4 ounces orange juice with calcium for 12 weeks. We started with 1gm then increased the next day by a gram to reach the 4gm dose.
  Intervention group participants completed Project FUN (8 module online nutrition and physical activity program) individually (password protected) in the school computer lab along with a workbook also used to check intervention completion.
  Interventions: Dietary Supplement: Beneo Synergy 1; Behavioral: Project FUN
- Control (No Intervention): The control group participated in usual school activities only completing pre and post measures.

INTERVENTIONS:
Dietary Supplement: Beneo Synergy 1
  Other Names: oligofructose enhanced inulin
  Arms: Intervention
Behavioral: Project FUN — Project FUN, a culturally tailored online nutrition and physical activity program is based on the Health Promotion/ Transtheoretical Model. It includes 8 modules offered in a password-protected learning management system along with a workbook also used to assure intervention completion.
  Arms: Intervention

SUMMARY:
The purpose of this study was to determine the feasibility, acceptability, and initial efficacy of combining prebiotic (Beneo Synergy 1) and calcium treatment with Project FUN (an online nutrition and physical activity program) on body composition and intestinal microbiota among 4th and 5th grade children whose social determinants placed them at higher risk for obesity. This aim was addressed through testing the following hypotheses:

H1 Prebiotic and calcium supplementation in combination with Project FUN, will result in improved body composition scores, dietary fat percentage, and physical activity compared to a usual class control who did not receive the intervention.

H2 Higher counts of Bacteroides and Bifidobacterium as well as fewer Firmicutes in the stool samples will correlate with improvement in body composition scores.

Since this was a pilot community-based efficacy study, the following feasibility, acceptability, and descriptive research questions were also addressed:

RQ1 What percentages of participants submit stool samples, body composition assessments and complete at least 70 percent of the intervention over the course of a 12-week study? RQ2 What is the relationship between changes in body composition scores, dietary fat percentage, physical activity and microbiota in stool samples before and after the 12-week intervention?

DETAILED DESCRIPTION:
The purpose of this study was to determine the feasibility, acceptability, and initial efficacy of combining prebiotic (Beneo Synergy 1) and calcium treatment with Project FUN (an online nutrition and physical activity program) on body composition and intestinal microbiota among 4th and 5th grade children whose social determinants placed them at higher risk for obesity. This aim was addressed through testing the following hypotheses:

H1 Prebiotic and calcium supplementation in combination with Project FUN, will result in improved body composition scores, dietary fat percentage, and physical activity compared to a usual class control who did not receive the intervention.

H2 Higher counts of Bacteroides and Bifidobacterium as well as fewer Firmicutes in the stool samples will correlate with improvement in body composition scores.

Since this was a pilot community-based efficacy study, the following feasibility, acceptability, and descriptive research questions were also addressed:

RQ1 What percentages of participants submit stool samples, body composition assessments and complete at least 70 percent of the intervention over the course of a 12-week study? RQ2 What is the relationship between changes in body composition scores, dietary fat percentage, physical activity and microbiota in stool samples before and after the 12-week intervention? The sample included 4th- 5th grade students at two private urban schools where 98% were eligible for free or reduced fee lunch. Of the 123 consenting 56% were male; 71% Latinx; 15% African American; 14% Other. Three percent were underweight; 49% normal weight; 22% overweight; 25% obese.

Consenting Latinx (n=20) and African American (n=8) participants completed microbiome analysis. Of these 54% were male; 6.5% underweight; 38.7% normal weight; 32.3% overweight; 2.6% obese.

ELIGIBILITY:
Inclusion Criteria:

* 4th- 5th grade students at two private urban schools where 98% were eligible for free or reduced fee lunch.

Exclusion Criteria:

* Parents indicated their child had taken an antibiotic in the last month since antibiotics can change intestinal flora though none required exclusion for this reason or for illness preventing participation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2012-11-13 (Actual); Primary Completion 2013-04-11 (Actual); Study Completion 2013-04-11 (Actual)

PRIMARY OUTCOMES:
Body mass index percentile mean change from baseline after 12 weeks | Pre and after 12-week intervention
  Weights to the nearest tenth of a pound were collected using a Seca model 8761321004 scale. Heights in stocking feet were measured to the nearest hundredth of an inch with a stadiometer (Seca Model 213, Hanover, MD, USA). Body mass index percentile was calculated using the Centers for Disease Control and Prevention school algorithm including birth date, measurement date, height, and weight

SECONDARY OUTCOMES:
Body fat percentage mean change from baseline after 12 weeks | Pre and after 12-week intervention
  Measured with the Omron HBF-306C hand-held bioimpedance monitor
Gut microbiota mean change from baseline after 12 weeks (Intervention group only) | Pre and after 12-week intervention
  Genomic markers of stool samples were analyzed by Roche 454 pyrosequencing of fecal 16S rDNA and validated by quantitative polymerase chain reaction.

OTHER OUTCOMES:
Dietary fat percentage mean change from baseline after 12 weeks | Pre and after 12-week intervention
  A 21-item, five-option response format measure was used developed by Prochaska JJ, Sallis JF, Rupp J. Screening measure for assessing dietary fat intake among adolescents.
Physical activity mean change from baseline after 12 weeks | Pre and after 12-week intervention
  Prochaska JJ, Sallis JF, Long B. A physical activity screening measure for use with adolescents in primary care.

IPD SHARING:
Plan to Share IPD: No
At this time there is no data repository for sharing of individual data.